CLINICAL TRIAL: NCT05873348
Title: A Controlled Study on Regulation of Systemic Inflammation by Fecal Bacteria Transplantation in Patients With COVID-19.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Huanlong Qin, chief physician, Shanghai 10th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMT-COVID-19-230207
Record Dates: First submitted 2023-05-23; First posted 2023-05-24 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Fecal Microbiota Transplantation; COVID-19 Infection
MeSH Terms: conditions — COVID-19 | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMTgroup (Experimental)
  Interventions: Procedure: Fecal microbiota transplantation
- control gtoup (No Intervention)

INTERVENTIONS:
Procedure: Fecal microbiota transplantation — Fecal microbiota transplantation (FMT) is the use of functional microorganisms in the feces of healthy people to form capsules and orally administer them to the intestinal tract of patients to reconstruct the intestinal flora of patients, so as to achieve the purpose of treating intestinal and exenteric diseases.
  Arms: FMTgroup

SUMMARY:
A total of 30 hospitalized patients with COVID-19 over 60 years old were enrolled in this study and were divided into the experimental group (n=15) and the control group (n=15) at a ratio of 1:1. Both groups were treated according to the 2022 Shanghai guidelines for Diagnosis and Treatment of COVID-19 infection and the hierarchical diagnosis and treatment process. The experimental group was treated with fecal microbiota transplantation (FMT) capsules for 1 week, and the control group was treated with empty capsules. Patients in both groups were followed up for 1 month after discharge. To observe the effect of combined FMT capsule treatment on the regulation of inflammatory factors in peripheral blood and the remodeling of intestinal flora, and to verify its safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Over 60 years old, male or female;

  2. Meet the diagnostic criteria of COVID-19;

  3. The patient signed the informed consent, agreed to receive FMT capsule treatment, agreed to cooperate with the whole process of the clinical trial, and agreed to collect clinical data and blood, saliva, urine, stool and other samples;

  4. The patient was able to swallow 3# capsules by herself.

Exclusion Criteria:

* 1. Confirmed diagnosis of non-COVID19 pneumonia;

  2. Critically ill patients requiring mechanical ventilation, or patients who are unable to eat by mouth and swallow 3# capsules;

  3. Patients who had undergone gastrointestinal surgery;

  4. Presence of intestinal organic lesions such as congenital megacolon, intestinal obstruction, intussusception, etc.

  5. Pathological intestinal inflammatory changes, such as inflammatory bowel disease;

  6. Planned use of antacids, probiotics, antibiotics, FMT and other treatments affecting intestinal flora within the past 3 months or the following 2 months;

  7. Patients and their families did not agree to receive FMT treatment;

  8. Patients unable to cooperate with follow-up visits.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Changes of inflammatory factors in the two groups | 7day,1month
  The changes of inflammatory factors in the transplantation group were detected compared with the control group

CONTACTS AND LOCATIONS:
Overall Officials: Long Li, Principal Investigator — Intestinal Microenvironment Treatment Center of General Surgery, Shanghai Tenth People's Hospital, Tenth People's Hospital of Tongji University
Locations (1):
- Li Long, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided